CLINICAL TRIAL: NCT01496807
Title: A Phase Ib Study of Yervoy With Sylatron for Patients With Unresectable Stages IIIB/C/IV Melanoma
Brief Title: Yervoy With Sylatron Unresectable Stage 3 or 4 Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16755
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-01

CONDITIONS: Melanoma
Keywords: unresectable; stage 3; stage 4; autoimmune; antibodies
MeSH Terms: conditions — Melanoma | interventions — peginterferon alfa-2b; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Yervoy with Sylatron (Experimental): Participants are given Yervoy induction every 3 weeks for four doses, for 12 weeks, and all participants simultaneously receive Sylatron induction weekly, followed by Sylatron maintenance alone for up to 144 additional weeks (total 156 weeks = 3 years).
  Interventions: Drug: Sylatron; Drug: Yervoy

INTERVENTIONS:
Drug: Sylatron — Sylatron - Once per week for 12 weeks, given as an injection under the skin.
  Other Names: PEG-Intron
Drug: Yervoy — Yervoy - Once every 3 weeks for 12 weeks (4 times total), given over a 90-minute intravenous infusion (through the vein).
  Other Names: Ipilimumab

SUMMARY:
The purpose of this study is to see how much of the drug Yervoy can be safely tolerated when it is given to people who are also receiving a drug called Sylatron. Investigators also wish to find out whether the addition of Yervoy increases the chance that Sylatron will cause a rise in the level of antibodies in the patient's blood that recognize their own tissues, known as "autoimmune" antibodies. Investigators also want to find out how likely it is that their tumor will shrink.

ELIGIBILITY:
Inclusion Criteria:

* Must have cytologically or histologically-confirmed and unresectable melanoma, previously untreated systemically other than a BRAF inhibitor for metastatic disease, meeting one of the following American Joint Committee on Cancer (AJCC) staging criteria: AJCC Stage IV (Tany,Nany,M1); AJCC Stage IIIB/C patients with unresectable nodal/locoregional involvement; Patients with cutaneous, ocular or mucosal melanoma are eligible
* Must have adequate hepatic, renal and bone marrow function as defined by the following parameters obtained within 4 weeks prior to initiation of study treatment. Hematologic Criteria: white blood count (WBC) >/= 3.0 x 10^9/L, Platelet > 100 x 10^9/L, Hemoglobin >/= 9 g/dL or 5.6 mmol/L; Renal and Hepatic Functional Criteria: Serum creatinine < 2.0 mg/dL or < 140 μmol/L, serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) < 2 times upper normal limit of laboratory normal (ULN)
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Must give informed consent according to institutional policy
* Must be willing to give written informed consent and must be able to adhere to dose and visit schedules
* Female patients of childbearing potential must be using a medically accepted method of birth control prior to Screening and agree to continue its use during the study or be surgically sterilized (e.g., hysterectomy or tubal ligation). Females of childbearing potential should be counseled in the appropriate use of birth control while in this study. Females who are not currently sexually active must agree and consent to use one of the above-mentioned methods should they become sexually active while participating in the study.
* Female patients of childbearing potential must have a negative serum pregnancy test (beta-hCG) at Screening.

Exclusion Criteria:

* Female patients who are pregnant, intend to become pregnant, or are nursing
* Previously treated with interferon alpha 2b, Sylatron or Yervoy therapy for melanoma
* Patients whose disease can be completely surgically resected
* Have not recovered from the effects of recent surgery
* Patients with a history of prior malignancy within the past 2 years other than surgically cured squamous or basal cell carcinoma of the skin, or cervical carcinoma in situ
* Have severe cardiovascular disease, i.e., arrhythmias requiring chronic treatment, congestive heart failure (NYHA Class III or IV) or symptomatic ischemic heart disease
* Patients with thyroid dysfunction not responsive to therapy
* Patients who, in the opinion of the investigator, have uncontrolled diabetes mellitus
* Suffering from an active autoimmune disease except medically controlled hypothyroidism and vitiligo
* An active and/or uncontrolled infection, including active hepatitis
* Have a history of seropositivity for HIV
* Pre-existing psychiatric condition, including but not limited to: History of severe depression (including Hospitalization for depression, Electroconvulsive therapy for depression, Depression that resulted in a prolonged absence from work and/or significant disruption of daily functions); Suicidal of homicidal ideation and/or suicidal or homicidal attempt; History of severe psychiatric disorders (e.g., psychosis, post-traumatic stress disorder or mania); Past history or current use of lithium and/or antipsychotic drugs
* A clinical diagnosis of substance abuse of the one or more of the following drugs, within the following timeframes, (not including time spent in detoxification, hospitalization or incarceration): Alcohol, intravenous drug use (IVDU), inhalational, psychotropics, narcotics, cocaine, prescription or over-the-counter drugs: within 1 year of the Screening visit; Receiving methadone, buprenorphine hydrochloride (HCL), and/or butorphanol tartrate within 1 year of Screening visit, unless participant has drug screen negative for other (non-narcotic) drugs documented in past year and repeated negative within 2 months of Screening visit; Multi-drug abuse (2 or more substances in 17a and 17b) within 3 years of Screening visit; If the patient's historic marijuana use is deemed excessive by the principal investigator (PI), or medically qualified individual or is interfering with the patient's life, then the patient is not eligible and should not be screened. If patient's marijuana use is not deemed excessive by PI and does not interfere with life, the patient must be instructed to discontinue any current use of recreational marijuana prior to entry into study.
* Patients with a medical condition requiring chronic systemic corticosteroids
* Known to be allergic to the drug substance or any of the excipients in the Sylatron or Yervoy formulation
* Patients who are in a situation or have any condition that, in the opinion of the investigator, may interfere with optimal participation in the study
* Have used any investigational drugs within 30 days of study entry
* Are participating in any other clinical treatment study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-02-17; Primary Completion 2016-03-16 (Actual); Study Completion 2016-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Brohl, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Brohl AS, Khushalani NI, Eroglu Z, Markowitz J, Thapa R, Chen YA, Kudchadkar R, Weber JS. A phase IB study of ipilimumab with peginterferon alfa-2b in patients with unresectable melanoma. J Immunother Cancer. 2016 Dec 20;4:85. doi: 10.1186/s40425-016-0194-1. eCollection 2016. PMID 28031816
- See also: A phase IB study of ipilimumab with peginterferon alfa-2b in patients with unresectable melanoma — http://www.readcube.com/articles/10.1186/s40425-016-0194-1?author_access_token=q4OsayXrovStniJBXf5KJW_BpE1tBhCbnbw3BuzI2RPgg2JIGHBI3V3-ffseGUyjAuw9rUiDlEJbtg5ZLnbOf6_A1R3uJM6OsFjtrfI8OCUCx0vfNVtKTA0zp40r-hd7eg9LOaU91RAq_c6MepNx4Q%3D%3D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 17, 2012 and December 5, 2013, 33 patients were screened and 31 patients were enrolled on treatment at Moffitt Cancer Center.
Period: Overall Study
Arm/Group | Yervoy With Sylatron
Started | 31
Completed | 1
Not Completed | 30
Not completed — Progressive Disease | 21
Not completed — Participant preference/toxicity | 8
Not completed — Change in diagnosis | 1

BASELINE CHARACTERISTICS:
Population: All evaluable participants will be those who completed treatment per study criteria.
Arm/Group | Yervoy With Sylatron
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 17
Age, Continuous [Median (Full Range); unit: years] | 65 [38 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Sylatron
Description: MTD of peginterferon alfa-2b (Sylatron) combined with Ipilimumab (Yervoy).
Time Frame: Up to 48 Months
Population: All participants
Measure: Number; unit: μg/kg s
Arm/Group | Yervoy With Sylatron
Number analyzed (Participants) | 31
μg/kg s | 2

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Ipilimumab
Description: MTD of Ipilimumab (Yervoy) combined with peginterferon alfa-2b (Sylatron). To assess the safety, toxicities and tolerability of a regimen of 3 μg/kg weekly Sylatron with concurrent induction Yervoy at 3 mg/kg, then if well tolerated, at 10 mg/kg every three weeks four times, in participants with unresectable stages IIIC/IV melanoma, and to define a well tolerated dose of Yervoy in that combination.
Time Frame: Up to 48 Months
Population: All participants
Measure: Number; unit: mg/kg
Arm/Group | Yervoy With Sylatron
Number analyzed (Participants) | 31
mg/kg | 3

3. Secondary Outcome: Number of Participants With Overall Response (OR)
Description: Overall Response: Complete Response (CR) + Partial Response (PR) by immune-related response criteria (irRC). Immune Related CR (irCR): Complete disappearance of all lesions (whether measurable or not, and no new lesions, and confirmation by a repeat consecutive assessment no less than 4 weeks from date first documented. Immure Related PR (irPR): decrease in tumor burden >50% relative to baseline confirmed by repeat consecutive assessment at least 4 weeks later.
Time Frame: Up to 54 Months
Population: All evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | Yervoy With Sylatron
Number analyzed (Participants) | 30
Participants
  Complete Response | 1
  Partial Response | 11

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Immune Related Progressive Disease (irPD): increase in tumor burden >25% relative to nadir (minimum recorded tumor burden) confirmed by repeat consecutive assessment at least 4 weeks later.
Time Frame: Up to 54 Months
Population: All evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Yervoy With Sylatron
Number analyzed (Participants) | 30
months | 5.9 [2.8 to 11.2]

5. Secondary Outcome: Overall Survival (OS)
Description: OS: The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive.
Time Frame: Up to 54 Months
Population: All evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Yervoy With Sylatron
Number analyzed (Participants) | 30
months | NA [29.5 to NA] — NA: The median overall survival was not reached in this study, with 18 patients (60%) alive at the time of censoring with a median follow-up of 35.8 months (range 19.7-50.2 months).

6. Secondary Outcome: Treatment Related Adverse Events (AEs) - Grade 3 to 5
Description: Percentage of participants with treatment related AEs, Grade 3 to 5. All adverse events, regardless of causality are also reported in the Serious Adverse Event/Other Adverse Event reporting area.
Time Frame: 4 Years, 1 Month
Population: All Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Yervoy With Sylatron
Number analyzed (Participants) | 31
Participants
  Grade 3 Adverse Events | 15
  Grade 4 Adverse Events | 0
  Grade 5 Adverse Events | 0
  None Reported | 16

7. Other Pre Specified Outcome: Count of Participants Developing Positive Autoantibody Screen
Description: Number of participants who developed a positive result during treatment for one or more antibodies of a previously negative screen.
  This study was not designed to statistically test the efficacy of treatment, and no inferential analyses will be performed. Investigators planned to look for evidence of serologic and clinical autoimmunity.
Time Frame: Up to 54 Months
Population: All evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | Yervoy With Sylatron
Number analyzed (Participants) | 30
Participants | 12

ADVERSE EVENTS:
Time Frame: 4 years, 1 month
Arm/Group | Yervoy With Sylatron
Serious Adverse Events (participants affected / at risk) | 14/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yervoy With Sylatron (N=31)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Endocrine disorders - Other, hypopituitarism (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2)
Blurred vision (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 5 (5)
Death NOS (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Pain (General disorders) | 2 (3)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Central nervous system necrosis (Nervous system disorders) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, Paresthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yervoy With Sylatron (N=31)
Fatigue (General disorders) | 29 (50)
Chills (General disorders) | 19 (24)
Fever (General disorders) | 15 (23)
General disorders and administration site conditions - Other, Intermittent bleeding of gums (General disorders) | 12 (18)
General disorders and administration site conditions - Other, Increased appetite (General disorders) | 12 (18)
General disorders and administration site conditions - Other, Decreased appetite (General disorders) | 12 (18)
General disorders and administration site conditions - Other, Occasional chest tightness (General disorders) | 12 (18)
General disorders and administration site conditions - Other, Leg cramps (General disorders) | 12 (18)
General disorders and administration site conditions - Other, Cold sweats (General disorders) | 12 (18)
Flu like symptoms (General disorders) | 8 (9)
Injection site reaction (General disorders) | 7 (7)
Pain (General disorders) | 6 (8)
Infusion related reaction (General disorders) | 3 (3)
Malaise (General disorders) | 3 (4)
Non-cardiac chest pain (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 19 (36)
Diarrhea (Gastrointestinal disorders) | 18 (41)
Constipation (Gastrointestinal disorders) | 12 (13)
Vomiting (Gastrointestinal disorders) | 10 (17)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Dry mouth (Gastrointestinal disorders) | 5 (6)
Gastrointestinal disorders - Other, Mouth sores (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (3)
Flatulence (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 26 (42)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 23 (45)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 8 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (5)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (9)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 3 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 19 (30)
Dizziness (Nervous system disorders) | 9 (10)
Dysgeusia (Nervous system disorders) | 9 (9)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 17 (21)
Dehydration (Metabolism and nutrition disorders) | 4 (5)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (6)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (5)
White blood cell decreased (Investigations) | 10 (26)
Alanine aminotransferase increased (Investigations) | 8 (9)
Aspartate aminotransferase increased (Investigations) | 8 (9)
Neutrophil count decreased (Investigations) | 6 (16)
Platelet count decreased (Investigations) | 6 (10)
Lymphocyte count decreased (Investigations) | 5 (14)
Weight loss (Investigations) | 5 (5)
Alkaline phosphatase increased (Investigations) | 2 (3)
Creatinine increased (Investigations) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal and connective tissue disorder - Other, Temporomandibular joint pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal and connective tissue disorder - Other, Muscle spasms, Left side (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (14)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Eye disorders - Other, Visual disturbance (Eye disorders) | 2 (2)
Eye disorders - Other, Double vision (Eye disorders) | 2 (2)
Eye disorders - Other, specify (Eye disorders) | 7 (9)
Blurred vision (Eye disorders) | 3 (3)
Dry eye (Eye disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 6 (7)
Depression (Psychiatric disorders) | 6 (8)
Confusion (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Endocrine disorders - Other, Night sweats (Endocrine disorders) | 4 (6)
Anemia (Blood and lymphatic system disorders) | 6 (15)
Hearing impaired (Ear and labyrinth disorders) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 3 (3)
Urinary tract infection (Infections and infestations) | 4 (9)
Hypertension (Vascular disorders) | 3 (6)
Hot flashes (Vascular disorders) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes